CLINICAL TRIAL: NCT03292523
Title: Work Productivity in Hyperventilation Syndrome
Acronym: WHY
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2016_68; 2017-A01542-51 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2017-09-21; First posted 2017-09-25 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Hyperventilation Syndrome
Keywords: Hyperventilation syndrome; Work productivity; Absenteeism; Presenteeism
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hyperventilation syndrome
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — Work Productivity and Activity Impairment (WPAI) Multidimensional Dyspnea Profile (MDP) Baseline Dyspnea Index (BDI), MOS-SF36, Hospital Anxiety Depression (HAD) Cognitive Failure Questionnaire (CFQ).

SUMMARY:
Hyperventilation syndrome is associated with impaired quality of life. The aim of the study is to assess the relationship between work productivity, including absenteeism and presenteeism, and the severity of hyperventilation syndrome

ELIGIBILITY:
Inclusion Criteria:

* Holders of employment contracts for at least 8 days
* Diagnosis of hyperventilation syndrome confirmed by:

Compatible symptoms and at least two symptoms reproduced by the hyperventilation challenge test: Nijmegen's score> 23 ; Demonstration of alveolar hyperventilation ( Either on rest blood and / or at rest (PaCO2 at rest <36 mmHg and D (A-a) O2 normal; Either during the HV test (increased recovery time of the basic PETCO2 after voluntary hyperventilation (greater than 5 minutes)

Exclusion Criteria:

* Existence of another chronic pulmonary disease (asthma, bronchial dilation, COPD, diffuse interstitial pneumonia, neuromuscular pathology ...) or cardiac (rhythm disorder, ischemic heart disease ...) which can participate in dyspnea
* Psychiatric illness / psychotropic treatment
* Pregnancy
* Patient already included in a clinical research protocol involving new therapeutics may not be included in this protocol
* Specific physiotherapy or previous training

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with confirmed hyperventilation syndrome, virgin of any treatment.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2021-02-23 (Actual); Study Completion 2021-02-23 (Actual)

PRIMARY OUTCOMES:
Association between the WPAI score and the Nijmegen score | At the time of diagnosis (Baseline)

SECONDARY OUTCOMES:
Association between the WPAI score and dyspnea scales | At the time of diagnosis (Baseline)
Association between the WPAI score and quality of life scores | At the time of diagnosis (Baseline)
Association between the WPAI score and PaCO2 | At the time of diagnosis (Baseline)
Association between the WPAI score and the Cognitive Failure Questionnaire score | At the time of diagnosis (Baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Cécile Chenivesse, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Calmette,CHU, Lille, France